CLINICAL TRIAL: NCT05070520
Title: Efficacy of Antimalarial Drugs Used for the Treatment of Uncomplicated Malaria, Plasmodium Falciparum, at the Agadez, Gaya and Tessaoua Sentinel Sites
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Programme National de Lutte contre le Paludisme, Niger (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 033/2020/CNERS
Record Dates: First submitted 2021-09-24; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: MALARIA
Keywords: Malaria; Efficacy; Arthemeter; Lumefantrine; Niger
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: This surveillance study is a prospective one-arm evaluation of clinical and parasitological responses to treatment of uncomplicated malaria with direct observation of treatment. Individuals with uncomplicated malaria, who meet the study inclusion criteria, will be recruited and treated at the sites by AL. They will be monitored for 28 days. Follow-up will consist of a series of fixed-date monitoring visits and corresponding clinical examinations and laboratory tests. Based on the results of these assessments, patients will be classified as having treatment failure (early or late) or adequate response. The proportion of patients with treatment failure during follow-up will be used to assess the efficacy of the study drugs.
  PCR analysis will be used to distinguish between true recrudescence due to treatment failure and episodes of re-infestation. A proportion of 10% of the slides read in the field will be submitted for quality control.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Artemether-lumefantrine — Efficacy of artemether lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria in three sentinel sites in Niger (Agadez, Gaya and Tessaoua) in 2020

SUMMARY:
In Niger, malaria is a major public health problem. It is the main cause of morbidity and mortality among children. The management of malaria cases is based on the principle of early diagnosis and rapid treatment with effective drugs. It is confronted with the appearance of strains resistant to antimalarial drugs, hence the need to monitor antimalarial drug sensitivity.

The study was conducted in three regions representing epidemiological strata of the country: Agadez (Centre de santé Intégré of Dagamanet in the Health district of Agadez), Maradi (Centre de santé intégré of Guindaoua in Tessaoua) and Dosso (Centre de santé Intégré centre in Gaya). The protocol used is the WHO standardized protocol of 2009. Artemether/Lumefantrine (AL) was administered with a 28-day follow-up in children aged 3 months to 15 years. A Polymerase Chain Reaction (PCR) correction is planned to differentiate between treatment failure and re-infestation as well as a study of genes responsible for resistance on the main drugs used.

DETAILED DESCRIPTION:
The study took place from September 1 to October 31, 2020 at the time of peak malaria transmission. It took place at three sentinel sites of the National Malaria Control Program (NMCP). These were in the regions of i) Agadez at the Centre de Santé Intégré (CSI) of Dagamanet in the Agadez district, ii) Dosso at the CSI centre in the health district (HD) of Gaya iii) Maradi at the CSI Guindaoua in the HD of Tessaoua. These sites were identified by the NMCP because of their high attendance rate and belong to 3 different malaria epidemiological strata.

As the treatment failure rate of artemether lumefantrine (AL) in the regions is unknown, 5% was chosen. With a confidence level of 95% and a precision around the estimate of 5%, a minimum of 73 patients were included. The number of patients was increased by 20% to account for possible dropouts and withdrawals during the 28/42 day follow-up period, 88 patients were included in the study per site.

The study drug is oral AL. It is one of the four antimalarial drugs selected by the Niger's NMCP for the management of malaria. The product consists of blister packs of 6 tablets, box of 30 of lot number K U142 with an expiration date of January 2022 and blister packs of 12 tablets, box of 30 of lot number K U456 with an expiration date of January 2022.

The AL combination was administered at a dose of 4 mg artemether and 24 mg lumefantrine per kg for three days. The AL was provided by the NMCP.

The different prescriptions were as follows:

* 5 to 15 Kg: 1 tablet, twice a day for three days.
* 15 to 25 Kg: 2 tablets, twice a day for three days.
* 25 to 35 kg: 3 tablets, twice a day for three days.
* Over 35 kg: 4 tablets, twice a day for three days.

The first day's intake was done under direct observation and possible side effects were noted. Any patient who persistently vomited after taking the medication was excluded from the study and treated with artesunate. Patients were followed up regularly until Day 28 and received a clinical examination with thick drop control and axillary temperature taking at Day 0, Day 1, Day 2, Day 3, Day 7, Day 14, Day 21, and Day 28. Capillary blood on filtered paper (Wattman) was routinely collected from all patients on the day of inclusion ( Day 0) and during follow-up for molecular analysis. For follow-up, the density of asexual parasite forms was assessed on the basis of 8 000 leukocytes per microliter of blood. All slides were read by two microscopists to ensure control. At the end of the follow-up, the response to treatment was classified according to clinical and parasitological criteria

ELIGIBILITY:
Inclusion Criteria:

* Brachial circumference (BC) > 125 mm and P/T z-score > -2 Standard Deviation (SD)
* Age between three months and fifteen years,
* Monospecific Plasmodium falciparum infestation detected by microscopy;
* Parasitemia between 1000 and 200000 asexual parasitic forms/µl ;
* Axillary temperature ≥37.5° or history of fever in the past 24 hours ;
* Ability to take oral medications;
* Ability and willingness to adhere to the protocol for the duration of the study and to adhere to the visit schedule ;
* Informed consent of the accompanying person (guardian or parent).

Exclusion Criteria:

* Inability to take oral medications
* History of antimalarial treatment in the past two weeks, including sulfadoxine-pyrimethamine (SPAQ) for seasonal malaria chemoprevention (SMC)
* Lack of consent for pregnancy testing
* Presence of general danger signs in children under five years of age or signs of severe P. falciparum malaria as defined by World Health Organization (WHO);
* Mixed infestation or monospecific infestation with another Plasmodium species, detected by microscopic examination;
* Severe malnutrition defined by a BC <125 mm AND P/T z-score < -3 Standard Deviation (SD)
* Moderate malnutrition defined by a BC <125 mm AND a -3 ≤P/T z-score < -2 SD
* Febrile condition due to illnesses other than malaria (e.g., measles, acute lower respiratory tract infection, severe diarrheal illness with dehydration) or other known chronic or severe underlying illnesses (e.g., cardiac, renal, or liver disease, HIV/AIDS) ;
* Regular use of medications that may interfere with antimalarial pharmacokinetics;
* History of hypersensitivity or contraindication to any of the drugs tested or used as replacement therapy;
* Lack of informed consent from the patient or accompanying person

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 259 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with asexual falciparum parasitaemia on Day 0. | 4 weeks
  Parasitaemia always refers to falciparum species. Mixed infections detected by light microscopy was excluded.
Number of patiants with presence of gametocytes on Day 0 | 4 weeks
Percentage of patients with danger signs of malaria on Day 1 | 4 weeks
  Depending on the classification, a patient will be considered as having experienced treatment failure if the danger signs are associated with the presence of parasites.
Proportion of patients with 'adequate clinical and parasitological response' (ACPR) before PCR-corrected | 8 weeks
  absence of parasitaemia on day 28 (day 42), irrespective of axillary temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure
Proportion of patients with 'adequate clinical and parasitological response' (ACPR) after PCR-corrected | 24 weeks
  PCR analysis
Proportion of patients with 'early treatment failure' (ETF) before PCR-corrected | 8 weeks
  * Danger signs or severe malaria on day 1, 2 or 3, in the presence of parasitaemia;
  * Parasitaemia on day 2 higher than on day 0, irrespective of axillary temperature;
  * Parasitaemia on day 3 with axillary temperature ≥ 37.5 °C; and
  * Parasitaemia on day 3 ≥ 25% of count on day 0
Proportion of patients with 'early treatment failure' (ETF) after PCR-corrected | 24 weeks
  -PCR analysis
Proportion of patients with 'late clinical failure' (LCF) before PCR-corrected | 8 weeks
  * danger signs or severe malaria in the presence of parasitaemia on any day between day 4 and day 28 (day 42) in patients who did not previously meet any of the criteria of early treatment failure; and
  * presence of parasitaemia on any day between day 4 and day 28 (day 42) with axillary temperature ≥ 37.5 °C in patients who did not previously meet any of the criteria of early treatment failure
Proportion of patients with 'late clinical failure' (LCF) after PCR-corrected | 24 weeks
  PCR analysis
Proportion of patients with 'late parasitological failure' (LPF) before PCR-corrected | 8 weeks
  presence of parasitaemia on any day between day 7 and day 28 (day 42) with axillary temperature < 37.5 °C in patients who did not previously meet any of the criteria of early treatment failure or late clinical failure.
Proportion of patients with 'late parasitological failure' (LPF) after PCR-corrected | 24 weeks
  PCR analysis
Percentage of the known mutations associated with artemisinin resistance observed. | 24 weeks
  PCR analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hadiza JACKOU, Dr, Principal Investigator — PROGRAMME NATIONAL DE LUTTE CONTRE LE PALUDISME
Locations (1):
- Programme National de Lutte Contre Le Paludisme, Niamey, Niger

IPD SHARING:
Plan to Share IPD: Undecided
Data could be used for thesis

REFERENCES:
- [Result] Severe falciparum malaria. World Health Organization, Communicable Diseases Cluster. Trans R Soc Trop Med Hyg. 2000 Apr;94 Suppl 1:S1-90. No abstract available. PMID 11103309
- [Derived] Laminou IM, Issa I, Adehossi E, Maman K, Jackou H, Coulibaly E, Tohon ZB, Ahmed J, Sanoussi E, Koko D. Therapeutic efficacy and tolerability of artemether-lumefantrine for uncomplicated Plasmodium falciparum malaria in Niger, 2020. Malar J. 2024 May 13;23(1):144. doi: 10.1186/s12936-024-04945-8. PMID 38741101